CLINICAL TRIAL: NCT02603068
Title: Multicenter, Randomized, Open Label Trial to Evaluate the Safety and Efficacy of Oral Treprostinil in Subjects With Pulmonary Hypertension Associated With Pulmonary Fibrosis
Brief Title: Oral Treprostinil in Subjects With Pulmonary Hypertension Associated With Pulmonary Fibrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study design was inadequate and would not achieve study endpoints
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-204
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Hypertension; Pulmonary Fibrosis
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Fibrosis | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Maximum Tolerated Dose (iMTD) (Experimental): Subjects are allowed to titrate oral treprostinil up to a maximum dose of 12 mg TID.
  Interventions: Drug: Oral treprostinil
- Fixed Dose (FD) (Experimental): Subjects are allowed to titrate oral treprostinil up to a maximum dose of 1 mg TID.
  Interventions: Drug: Oral treprostinil

INTERVENTIONS:
Drug: Oral treprostinil — Oral treprostinil will be administered as TID dosing for up to 16 Weeks.
  Other Names: Orenitram

SUMMARY:
This multicenter, randomized, open-label study will assess the safety and efficacy of oral treprostinil in subjects diagnosed with pulmonary hypertension associated with pulmonary fibrosis.

DETAILED DESCRIPTION:
This study will evaluate how oral treprostinil can affect pulmonary vascular resistance, as assessed by right heart catheterization, and exercise capacity, as assessed by the Six-Minute Walk Test. This is a 16-week study that will involve at least 10 clinical trial centers. The expected enrollment period is around 24 months and 52 subjects will be entered into the study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily gives informed consent
* Must meet criteria for lung transplant referral but is not required to be on an active lung transplant list
* Stable and significant diffuse parenchymal lung disease with a diagnosis of interstitial lung disease
* 6MWD greater than or equal to 75 meters
* Right heart catheterization with a mean pulmonary arterial pressure >= 30 mgHg, pulmonary capillary wedge pressure <= 15 mmHg and pulmonary vascular resistance > 240 dynes
* Echo-Doppler examination showing evidence of right ventricular dysfunction and normal left diastolic ventricular function
* Either not receiving any PAH-approved oral therapy, or is receiving monotherapy (ERA, PDE-5I, or riociguat) for > 60 days and receiving a stable dose for > 30 days prior to enrollment
* Able to communicate effectively with study personnel and will to be cooperative with protocol requirements

Exclusion Criteria:

* History of repaired or unrepaired congenital heart disease
* Received prostanoid therapy in the past 30 days, or has shown an intolerance or lack of efficacy to prostanoid therapy resulting in discontinuation or inability to titrate prostacyclins
* Diagnosis of sarcoidosis
* History of thromboembolic disease
* Chronic renal insufficiency
* Pregnancy or lactating
* Currently receiving an investigational drug, has an investigational device in place, or has participated in an investigational drug or device study within 30 days prior to Screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance (PVR) | Baseline to Week 16
  Change in PVR between iMTD and fixed dose groups

SECONDARY OUTCOMES:
Change in Six-minute walk distance (6MWD) | Baseline to Week 16
  Change in 6MWD between iMTD and fixed dose groups
Change in N-terminal pro-brain natriuretic peptide (NT-ProBNP) | Baseline to Week 16
  Change in NT-ProBNP between iMTD and fixed dose groups

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, MD, Principal Investigator — University of California, Los Angeles - Pulmonary Division
Locations (7):
- United States (7):
  - Banner University Medical Center Phoenix Advanced Lung Disease, Phoenix, Arizona
  - University of California, Los Angeles - Pulmonary Division, Los Angeles, California
  - University of California - Davis Medical Group, Sacramento, California
  - Emory University Hospital, Atlanta, Georgia
  - Johns Hopkins University, Baltiomore, Maryland
  - Oregon Health and Science University, Portland, Oregon
  - CLC Pulmonary Hypertension Clinic Division of Pulmonary, Allergy and Critical Care Medicine UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Study is withdrawn. There is no data to share.